CLINICAL TRIAL: NCT00709241
Title: Prognostic Value of Negative Affectivity in Patients With Heart Failure
Brief Title: Psychosocial Patterns and Prognosis in Patients With Heart Failure
Acronym: PANIC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P051044
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Systolic Heart Failure; Diastolic Heart Failure
Keywords: Heart failure; Psychosocial factors; Depression; Patient compliance
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure, Diastolic; Heart Failure; Depression; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine.
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective observational study is designed to confirm the prognostic and economic impact of depression in ambulatory patients with systolic or diastolic heart failure, to explore the impact of other psychosocial patterns such as type D personality, anxiety disorders, locus of control, perceived social support, anger, hopelessness, and to evaluate potential pathophysiological and behavioral pathways.

DETAILED DESCRIPTION:
Studies suggest that depressive symptoms may be associated with a worse prognosis and higher costs of care in patients with chronic heart failure in some populations, but such data in a French population are missing. On the other hand, little is known of the impact of other psychosocial dysfunction whereas the pathophysiology of this association remains hypothetical.

Main objective: to confirm the impact of depressive symptoms on cardiovascular death in ambulatory heart failure patients

Other objectives:

* to study the impact of depressive symptoms on sudden death, non cardiovascular death, and hospitalization rates;
* to study the role of other psychosocial patterns or personality traits such as anxiety disorders, locus of control, perceived social support, anger, hopelessness, optimism and type D personality in cardiovascular and total mortality;
* to study the interaction with patient behaviors (drug compliance, addictions);
* to explore some pathophysiological pathways (chronic inflammation and chronic loss of myocytes),
* and to evaluate the impact of psychosocial distress on health care costs. Design: multicenter observational study with a minimum of 2 year follow up Population: 700 ambulatory patients, aged above 18 y.o., with acute heart failure within the last 24 months

Methodology:

* psychosocial patterns and personality traits are assessed using validated self-administered questionnaire; use of the Beck Depression Index in this population is validated against the Montgomery & Asberg Depression Rating Scale evaluation
* cardiac condition is evaluated at pre-defined time period by B-natriuretic peptide levels, echocardiography and 6'-walk test

End-point criteria:

* primary : rate of cardiovascular death
* secondary : rate of total mortality and sudden death, rate of rehospitalization for heart failure and for any cause, total and specific health care costs.

ELIGIBILITY:
Inclusion Criteria:

* age above 18,
* acute heart failure within the last 24 months
* stable cardiovascular condition for at least 2 weeks
* non hospitalized, non institutionalized patient,
* french speaking and reading,

Exclusion Criteria:

* Non inclusion criteria :
* curable cardiomyopathy, cardiomyopathies associated with systemic illnesses (Lupus...), neurodegenerative or pulmonary illnesses, or hypertrophic/restrictive cardiomyopathy
* unstable cardiovascular condition
* heart transplant and hemodialysis patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2007-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | 2 years

SECONDARY OUTCOMES:
total mortality, sudden death rate, non cardiovascular mortality, rate of hospitalization, of rehospitalization for heart failure, of hospitalization for cardiovascular and non cardiovascular reasons,total health care costs and nature of theses costs | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: François LEDRU, MD PH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Georges pompidou, Paris, France